CLINICAL TRIAL: NCT03266354
Title: Changes of the Corneal Endothelial Cell Count After Artisan Phakic Intraocular Lens Implantation
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Omar, resident, Assiut University
Other Study IDs: CECCAPIOL
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-05

CONDITIONS: High Myopia
Keywords: Artisan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: specular microscopy before and after Artisan PIOL — specular microscopy will be performed before and after implantation of the rigid Artisan iris-fixated pIOL to analyze the change in corneal endothelial cell count

SUMMARY:
the investigator will evaluate the change in endothelial cell count in eyes implanted with the iris-claw phakic Artisan lens for treatment of moderate to high myopia using specular microscopy

DETAILED DESCRIPTION:
Iris-fixated phakic intraocular lenses (pIOLs) are used worldwide to correct high myopia, hyperopia, and astigmatism. It is used to correct high degrees of myopia in patients for whom laser excimer refractive surgery is not indicated.

The Artisan lens is designed to minimize the contact between the iris and the IOL resulting in less halo and glare from the prism effect.

Several clinical studies show that the visual results of the Artisan lens are stable and predictable. Artisan phakic IOLs provides precise predictability.

There have been concerns that the anterior chamber lens could damage the endothelial cell layer because of its proximity to the cornea. The manufacturer advises using the Artisan lens only in eyes with an ECD greater than 2000 cells/mm2 and an ACD greater than 2.6 mm.

Corneal endothelium is metabolically active and responsible for keeping the corneal stroma in its usual dehydrated state of 70% water.

loss of endothelial cells from increasing age, trauma, disease, or corneal surgery can reduce the density of endothelial cells and affect the ability of the endothelium to maintain it's primary function.

Alterations in the corneal endothelium depend on surgical technique and style; although endothelial cell loss is mainly the result of surgical trauma, continuous endothelial cell loss can occur. Late corneal decompensation often occurs in the absence of direct intraoperative endothelial trauma. These complications can be explained by the toxic effect of inflammatory mediators on the corneal endothelium.

Specular microscopy is used to view and record non-invasively the image of the corneal endothelial cell layer.

ELIGIBILITY:
Inclusion Criteria:

* an age greater than 20 years, stable myopia with a variation in spherical equivalent of less than -0.50 diopter (D) during the 12 month preoperative period, a normal anterior segment with an ACD (i.e., the area between the corneal endothelium and the central anterior lens capsule) greater than 3.00 mm, an endothelial cell count of 2000 cells/mm2 or greater, no corneal, pupil, or iris abnormalities; and no history of glaucoma and chronic or recurrent uveitis , having contraindications to laser in situ keratomileusis based on pachymetric data or other corneal shape characteristics, and an intraocular pressure of 20 mm Hg or less.

Exclusion Criteria:

* an ACD less than 3.0 mm, history of ocular surgery, glaucoma, chronic uveitis, or preexisting ocular pathologic features or abnormalities.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Artisan PIOL
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in the Corneal endothelial cell count after Artisan phakic intraocular lens implantation | 5 minutes
  specular microscopy will be performed on a number of myopic patients before and after implantation of the rigid Artisan iris-fixated pIOL to analyze the change in corneal endothelial cell count.

CONTACTS AND LOCATIONS:
Overall Officials: gamal rashed, professor, Study Chair — Assiut University
Locations (1):
- Fculty of medicine, Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Menezo JL, Peris-Martinez C, Cisneros AL, Martinez-Costa R. Phakic intraocular lenses to correct high myopia: Adatomed, Staar, and Artisan. J Cataract Refract Surg. 2004 Jan;30(1):33-44. doi: 10.1016/j.jcrs.2003.11.023. PMID 14967266
- [Background] Menezo JL, Avino JA, Cisneros A, Rodriguez-Salvador V, Martinez-Costa R. Iris claw phakic intraocular lens for high myopia. J Refract Surg. 1997 Sep-Oct;13(6):545-55. doi: 10.3928/1081-597X-19970901-11. PMID 9352483
- [Background] Menezo JL, Cisneros AL, Rodriguez-Salvador V. Endothelial study of iris-claw phakic lens: four year follow-up. J Cataract Refract Surg. 1998 Aug;24(8):1039-49. doi: 10.1016/s0886-3350(98)80096-5. PMID 9719962
- [Background] Benedetti S, Casamenti V, Benedetti M. Long-term endothelial changes in phakic eyes after Artisan intraocular lens implantation to correct myopia: five-year study. J Cataract Refract Surg. 2007 May;33(5):784-90. doi: 10.1016/j.jcrs.2007.01.037. PMID 17466848
- [Background] STOCKER FW. The endothelium of the cornea and its clinical implications. Trans Am Ophthalmol Soc. 1953;51:669-786. No abstract available. PMID 13216798
- [Background] Mishima S. Clinical investigations on the corneal endothelium. Ophthalmology. 1982 Jun;89(6):525-30. doi: 10.1016/s0161-6420(82)34755-7. PMID 6750487
- [Background] Waring GO 3rd, Bourne WM, Edelhauser HF, Kenyon KR. The corneal endothelium. Normal and pathologic structure and function. Ophthalmology. 1982 Jun;89(6):531-90. PMID 7122038
- [Background] Joyce NC. Cell cycle status in human corneal endothelium. Exp Eye Res. 2005 Dec;81(6):629-38. doi: 10.1016/j.exer.2005.06.012. Epub 2005 Jul 28. PMID 16054624
- [Background] Maurice DM. Cellular membrane activity in the corneal endothelium of the intact eye. Experientia. 1968 Nov 15;24(11):1094-5. doi: 10.1007/BF02147776. No abstract available. PMID 5721120
- [Background] Laing RA, Sandstrom MM, Leibowitz HM. In vivo photomicrography of the corneal endothelium. Arch Ophthalmol. 1975 Feb;93(2):143-5. doi: 10.1001/archopht.1975.01010020149013. PMID 1115675